CLINICAL TRIAL: NCT02412358
Title: Clinical Comparison of Three Types of Toothbrushes Pulsar, Crossaction and Butler on Gingivitis and Plaque Removal
Brief Title: Clinical Comparision of Three Types of Toothbrushes Pulsar, Crossaction and Butler on Gingivitis and Plaque Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Moeintaghavi, Professor of Periodontics, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 86394
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Healthy
Keywords: toothbrushing; plaque control; gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pulsar (Active Comparator): Patients use Pulsar toothbrush for plaque removal
  Interventions: Device: toothbrush
- Crossaction (Active Comparator): Patients use Crossaction toothbrush for plaque removal
  Interventions: Device: toothbrush
- Butler (Active Comparator): Patients use Butler toothbrush for plaque removal
  Interventions: Device: toothbrush

INTERVENTIONS:
Device: toothbrush
  Other Names: Pulsar, Crossaction, Butler toothbrush

SUMMARY:
* Objective: To compare clinical results of three types of manual tooth brushes on gingivitis and plaque removal efficacy.
* Material and Methods: This study is a single blind randomized trial with crossover design which involved 30 periodontally healthy individuals. At baseline professional plaque removal and oral hygiene instruction are performed for all the students, then they are asked to avoid brushing for 1-2 days. Thereafter plaque and gingivitis scores are measured using plaque and gingival indices (PI and GI). Then subjects are instructed to use Pulsar tooth brush for a two-week period and then, GI and PI indices are assessed again. After passing one-week period for wash out, subjects don't brush for 1-2 days and indices are recorded again. The same procedure are done for Cross action, and Butler 411 tooth brushes respectively.

DETAILED DESCRIPTION:
This study is a single blind randomized trial with crossover design which involved 30 periodontally healthy individuals. At baseline professional plaque removal and oral hygiene instruction are performed for all the students, then they are asked to avoid brushing for 1-2 days. Thereafter plaque and gingivitis scores are measured using plaque and gingival indices (PI and GI). Then subjects are instructed to use Pulsar tooth brush for a two-week period and then, GI and PI indices are assessed again. After passing one-week period for wash out, subjects don't brush for 1-2 days and indices are recorded again. The same procedure are done for Cross action, and Butler 411 tooth brushes respectively.

ELIGIBILITY:
Inclusion Criteria:

* having at least five teeth in each quadrant;
* no partial denture;
* no orthodontic banding or retention wires;
* no oral lesions or sites with probing pockets depth ≥ 5 mm;
* routine use of a manual toothbrush.

Exclusion Criteria:

* having any systematic disease which would influence the course of periodontal diseases or the response to the treatment
* smoking

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Plaque Index | 2 weeks
  it is an index used for scoring plaque accumulation
Gingival index | 2 weeks
  it is an index used for scoring gingival inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Amir Moeintaghavi, DDs., Msc., Principal Investigator — Mashhad University of Medical Sciences
Locations (1):
- Amir Moeintaghavi, Mashhad, Khorasan Razavi, Iran